CLINICAL TRIAL: NCT05999110
Title: Algarve Active Ageing - Cardiac and Osteoarthritis Rehabilitation: Personalized Physical Exercise Protocol in After Acute Myocardial Infarction or Cardiovascular Risk and Knee Osteoarthritis, a Randomized Controlled Trial
Brief Title: Algarve Active Ageing - Cardiac and Osteoarthritis Rehabilitation (A3-COR)
Acronym: A3-COR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associação para o Desenvolvimento do Centro Académico de Investigação e Formação Biomédica do Algarv (Network)
Collaborators: European Regional Development Fund (Other); Loulé Municipal Council (Unknown); Albufeira Municipal Council (Unknown); Quarteira Parish Council (Unknown)
Responsible Party: Principal Investigator, Sandra Rafael Pais, Researcher, Associação para o Desenvolvimento do Centro Académico de Investigação e Formação Biomédica do Algarv
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 072590 - A3-COR
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis, Knee; Myocardial Infarction, Acute; Hypertension; Dyslipidemias; Type 2 Diabetes; Smoking Habit
Keywords: Knee Osteoarthritis; Acute Myocardial Infarction; Cardiovascular Risk; Personalized Medicine; Healthy Ageing; Exercise; Personalized Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Myocardial Infarction; Hypertension; Dyslipidemias; Diabetes Mellitus, Type 2; Smoking; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are being assigned for two groups in parallel and a pre and post-test analysis is being performed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The participants receive twelve weeks of a supervised personalised exercise program, based on aerobic and strength training. This group also receives a behavioral change session with a psychologist and nutritional advice session with a nutritionist.
  Interventions: Other: Physical Exercise
- Control Group (No Intervention): This group receive no exercise intervention. The group receives equally as the exercise group, a behavioral change session with a psychologist and nutritional advice session with a nutritionist.

INTERVENTIONS:
Other: Physical Exercise — The intervention includes a personalized physical exercise program based on aerobic and strength training, with prior warm-up and post cool-down exercises. All participants also receive a nutritional advice session and a behavioral changes session.
  Arms: Exercise Group

SUMMARY:
This study aims to develop, implement, and determines the effectiveness of a personalized medicine approach to each individual's phenotype, based on an innovative physical exercise program to promote the treatment of pain and functional limitation resulting from knee osteoarthritis (KOA) in patients recovering after acute myocardial infarction (AMI) and cardiovascular risk (CVR).

This randomized clinical study is important due to the lack of evidence according to the effectiveness of a personalized physical exercise intervention in people after MI or CVR with simultaneous KOA.

Some studies have shown the existence of a relationship between OA and cardiovascular diseases (CVD), including coronary artery disease, stroke, congestive heart failure, peripheral arterial disease, cardiac procedures, or death related to CVD, since individuals with OA have a higher prevalence of CVD than individuals without OA.

Sedentary behaviour is a risk factor for AMI, CVR and KOA, and, at the same time, physical exercise is a common non-pharmacological treatment for people suffering from these conditions, namely in the control of joint pain, gains in functional capacity, and the improvement of cardiorespiratory functional capacity, whose impact can be felt in level of quality of life.

Chronic diseases have a significant impact on the global burden of disease, particularly CVD and OA, with the added presence of obesity also contributing to a high rate of all-cause morbidity and mortality, representing a substantial health burden and with growing implications for individuals, health systems and socioeconomic costs.

The presence of OA seems to lead to an increased risk of developing CVD. Several mechanisms have been proposed to explain this relationship. Chronic inflammation associated with OA is one of the hypotheses suggested to explain the increased risk of CVD in these individuals. Furthermore, the pain and disability associated with OA may also limit participation in exercise/physical activity, influencing other risk factors associated with both chronic diseases, such as weight gain.

The lack of studies about physical exercise intervention on people that suffered acute myocardial infarction or is in cardiovascular risk with simultaneous knee osteoarthritis and the lack of offer of phase III cardiac rehabilitation in Algarve motivated the development of this study, with the assumption of adopting a healthier lifestyle.

DETAILED DESCRIPTION:
A new exercise protocol (A3-COR Protocol) for patients with knee osteoarthritis (OA) recovering after acute myocardial infarction (AMI) or with cardiovascular risk (CVR) was developed and implemented. The purpose of the A3-COR protocol is to improve quality of life, functionality, and pain, through regular physical exercise facilitating an active and healthy lifestyle.

This clinical trial includes 2 parallel intervention groups with a pre- and post-test analysis. In the exercise group (EG), the participants will receive a twelve weeks of a supervised personalised exercise program and in the control group (CG) there will be no intervention. Both groups will have a behavioral change session with a psychologist to promote changes in lifestyle and a session with a nutritionist to promote healthy eating habits.

Both groups will be assessed two times, the pre-test in the beginning of the study (T0-Baseline) before starting the intervention or control and the post-test taking place at the end of 12 weeks (T1-Post-test).

The sample includes subjects from the community who met the defined eligibility criteria. Participation in the study is voluntary and sample recruitment will be carried out through publicity materials, such as flyers posted at senior universities, institutions/associations, municipalities, parish councils, sports complexes, health centres, among other public spaces of interest.

To calculate the sample size, the software G*Power was used. The primary outcome for this clinical trial was the knee-related pain, measured by the Knee Injury and Osteoarthritis Outcome Score (KOOS) with is a self-reported outcome with five subscales: 1) Symptoms+Stiffness; 2) Pain; 3) Function, daily living; 4) Function, sports and recreational activities and 5) Quality of Life, all score 0-100. According to the literature, an important clinical difference in the KOOS subscales has been suggested to be 8 to 10 points. Based on the expected difference of 10 points between the intervention and control groups and a standard deviation of 20 in Pain, 64 patients were required in each group with a significance level of 0.05 and power of 80%. With an estimated dropout rate of 10%, a total number of 142 subjects will be randomized to the EG (n = 71) and to the CG (n = 71).

The screening for acute myocardial infarction will be done with the presence of myocardial lesion detected by abnormal cardiac biomarkers evidencing acute myocardial ischemia. The screening of cardiovascular risk will consider the presence of any of the following cardiovascular risk factors: hypertension, dyslipidemia, or smoking habits, according to the SCORE2 or SCORE2 O.P. The screening of knee osteoarthritis will be done according to the National Institute for Health and Excellence (NICE) (2022)(NG226), EULAR evidence-based recommendations for the diagnosis of knee osteoarthritis (2009) and American College of Rheumatology (ACR)(1986) clinical criteria. To identify participants with cognitive impairment, the Montreal Cognitive Assessment (MoCA) instrument was applied and cutoff points for the Portuguese population considering age and educational level were used.

The training sessions combine cardiorespiratory exercises for the development of aerobic capacity and strength exercises, particularly resistant strength, in tasks that include open and closed chain exercises, using your own body weight and equipment for this purpose. The training zones are defined according to the performance of each individual in the test of cardiorespiratory fitness in effort and test of maximum isokinetic strength, carried out in the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older; Knee pain, Morning stiffness that lasts no longer than 30 minutes and one of the following: crepitus, restricted function, bony enlargement. Acute Myocardial Infarction with myocardial lesion detected by abnormal cardiac biomarkers evidencing acute myocardial ischemia; High risk level in the Systematic Coronary Risk Evaluation (SCORE2) or the Systematic Coronary Risk Evaluation Older Person (SCORE2 O.P.) cardiovascular risk algorithm or prior cardiovascular disease; Independent gait

Exclusion Criteria:

* Occurrence of acute myocardial infarction with less than 12 months; Cognitive impairment- Montreal Cognitive Assessment (MoCA); Type 1 diabetes or insulin dependence; Pacemaker device; Knee prosthesis; Currently doing formal exercise session for more that 30 minutes per week; Class III or IV angina according to Canadian Cardiovascular Society criteria; Class III or IV symptoms according to New York Heart Association criteria; Type 2 Myocardial Infarction; Uncontrolled and symptomatic cardiac arrythmia with hemodynamic impact; Severe and symptomatic aortic valve stenosis; Uncontrolled and symptomatic heart failure; Active myocarditis, pericarditis or endocarditis; Acute aortic syndrome; Known or suspected desiccant aneurism; Acute systemic infection.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Change the Level of Pain | 12 weeks
  Significant increase in pain subscore of Knee Injury and Osteoarthritis Outcome Score. The subscore can range between 0-100% and higher values mean less pain.
Change the Level of Function | 12 weeks
  Significant increase in both function subscores of Knee Injury and Osteoarthritis Outcome Score. The subscores can range between 0-100% and higher values mean better function.
Change the Time Up and Go Test Performance | 12 weeks
  Significant decrease in time (seconds) to perform the Timed Up and Go (TUG) test. Higher time of performance means poorer physical function.
Change the 30-Second Chair Stand Test Performance | 12 weeks
  Significant increase of number of repetitions in 30-second chair stand test. Higher number of repetitions in 30 seconds means better physical function.
Change the 40m Fast Paced Walk Test Performance | 12 weeks
  Significant decrease in time (seconds) of performance in 40m fast paced walk test. Higher time of performance means poorer physical function.
Change the Stair Climb Test Performance | 12 weeks
  Significant decrease in time (seconds) of performance in Stair Climb Test (9 steps). Higher time of performance means poorer physical function.
Change the 6 Minutes Walk Test Performance | 12 weeks
  Significant increase in distance (meters) in 6 Minutes Walk Test. Higher distance in 6 minutes means better physical function.
Change in Quality of Life | 12 weeks
  Significant increase in any subscore or total score of Medical Outcomes Study 36-item Short-Form Health Survey (SF-36), used to assess quality of life. Instrument can range between 0-100 and higher values mean better self-precepted quality of life.
Change in Peak Torque of Quadriceps and Hamstring Muscles | 12 weeks
  Significant increase in peak torque (N/m). Peak Torque of Quadriceps and Hamstring Muscles will be measured by a fixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Change in Work of Quadriceps and Hamstring Muscles | 12 weeks
  Significant increase in work per repetition (N/m). Work of Quadriceps and Hamstring Muscles will be measured by a fixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Change in Power of Quadriceps and Hamstring Muscles | 12 weeks
  Significant increase in power per repetition (N/m). Power of Quadriceps and Hamstring Muscles will be measured by a fixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Change in Peak torque time of Quadriceps and Hamstring Muscles | 12 weeks
  Significant increase in Peak torque time (s). Peak torque time of Quadriceps and Hamstring Muscles will be measured by a fixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Change in Force of Quadriceps and Hamstring Muscles | 12 weeks
  Significant increase in Force (kg). Force of Quadriceps and Hamstring Muscles will be measured by a fixed dynamometer with concentric/concentric action at an angular velocity of 60º per second for 5 repetitions of extension and flexion of each knee.
Change in Maximal Oxygen Uptake (VO2max) | 12 weeks
  Significant increase in Maximal Oxygen Uptake (VO2max). Higher VO2max means better cardiorespiratory function. The VO2max will be evaluated through the exercise cardiorespiratory test with progressive increase of the external load by the manipulation of the velocity or inclination.
Change in First Ventilatory Threshold (VT1 - VO2) | 12 weeks
  Significant increase in First Ventilatory Threshold (VT1 - VO2). Higher VT1 means better cardiorespiratory function. The VT1 will be evaluated through the exercise cardiorespiratory test with progressive increase of the external load by the manipulation of the velocity or inclination.
Change in Respiratory Compensation Point (RCP - VO2) | 12 weeks
  Significant increase in Respiratory Compensation Point (RCP - VO2). Higher RCP means better cardiorespiratory function. The RCP will be evaluated through the exercise cardiorespiratory test with progressive increase of the external load by the manipulation of the velocity or inclination.

SECONDARY OUTCOMES:
Change in maximal displacement of vastus lateralis and medialis, biceps femoris and semitendinous | 12 weeks
  Significant change maximal displacement (mm) of vastus lateralis and medialis, biceps femoris and semitendinous. Higher radial muscle belly displacement means poor muscle function and muscle atrophy. The muscle displacement will be measured by a tensiomyography system (TMG S2).
Change in contraction time of vastus lateralis and medialis, biceps femoris and semitendinous | 12 weeks
  Significant change in contraction time of vastus lateralis and medialis, biceps femoris and semitendinous. The contraction time will be measured by a tensiomyography system (TMG S2).
Change in Weight | 12 weeks
  Significant decrease in weight (kg). Higher values of weight mean poor body composition and health. The weight will be measured using bioimpedance.
Change in body mass index | 12 weeks
  Significant decrease in body mass index (kg/m2). Higher values of body mass index mean poor body composition and health. The body mass index will be measured using bioimpedance.
Change in fat mass | 12 weeks
  Significant decrease in fat mass (kg and %)). Higher values of fat mass mean poor body composition and health. The fat mass will be measured using the bioimpedance.
Change in fat-free mass | 12 weeks
  Significant increase in fat-free mass (kg and %). Higher values of fat-free mass mean better body composition and health. The fat-free mass will be measured using the bioimpedance.
Change in fat mass index | 12 weeks
  Significant decrease in fat mass index (kg/m2). Higher values of fat mass index mean poor body composition and health. The fat mass index will be measured using the bioimpedance.
Change in fat-free mass index | 12 weeks
  Significant increase in fat-free mass index (kg/m2). Higher values of fat-free mass index mean better body composition and health. The fat-free mass index will be measured using the bioimpedance.
Change in muscle mass index | 12 weeks
  Significant increase in muscle mass index (kg/m2). Higher values of muscle mass index mean better body composition and health. The muscle mass index will be measured using the bioimpedance.
Change in total body water | 12 weeks
  Significant increase in total body water (L and %). Higher values of total body water mean better body composition and health. The total body water will be measured using the bioimpedance.
Monitoring phase angle | 12 weeks
  Keep the phase angle within normal limits for the age. The phase angle will be measured using the bioimpedance.
Change in fat visceral fat | 12 weeks
  Significant decrease in visceral fat (L). Higher values of visceral fat mean poor body composition and health. The visceral fat will be measured using the bioimpedance.
Change in abdominal circumference | 12 weeks
  Significant decrease in abdominal circumference (cm). Higher values of abdominal circumference mean poor body composition and health. The abdominal circumference will be measured using measure tape, according to the STEPS Manual of the World Health Organization.
Change in Hand Grip Strength | 12 weeks
  Significant increase in hand grip strength (kg). Higher hand grip strength is correlated with higher functional status. Maximum handgrip strength will be measured with the Lafayette Digital and Dynamometer manual digital dynamometer on the dominant upper limb.
Change in Rescue's Pain Medication Posology | 12 weeks
  Decrease the necessity of rescue's pain medication related with knee osteoarthritis.
Change in hospital readmissions related to Myocardial Infarction | 12 weeks
  Decrease hospital readmissions related with Myocardial Infarction.
Change medical appointments number related with Myocardial Infarction | 12 weeks
  Reduce the number of appointments related with Myocardial Infarction.
Change medical appointments number related with Knee Osteoarthritis | 12 weeks
  Reduce the number of appointments related with Knee Osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra R Pais, PhD, Principal Investigator — AD-ABC
Locations (1):
- AD-ABC, Faro, Algarve, Portugal